CLINICAL TRIAL: NCT04904419
Title: Multi-center Research Project for Glioma Molecular Pathology Intraoperative Rapid Detection
Status: Completed | Type: Observational
Sponsor: Jinsong Wu (Other)
Responsible Party: Sponsor-Investigator, Jinsong Wu, Prof., Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: KY2020-1298
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Glioma, Malignant
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Intraoperative Rapid Detection mutation of IDH, TERT and BRAF v600e — Intraoperative Rapid Detection mutation of IDH, TERT and BRAF v600e

SUMMARY:
We explores the accuracy and sensitivity of rapid intraoperative detection of IDH, TERT, BRAF indicators through a prospective clinical multi-center study. This part includes a total of 300 fresh tissue samples, paired blood samples, relevant clinical information and follow-up information from 300 patients with different grades of adult glioma. By comparing with the postoperative sequencing results, the specificity and sensitivity of intraoperative IDH and TERT rapid detection results are clear.

ELIGIBILITY:
Inclusion Criteria:

* 1. Glioma patients with Informed Consent Form 2. Glioma patients with intact clinical information

Exclusion Criteria:

* 1. Glioma patients without Informed Consent Form 2. Glioma patients without intact clinical information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Glioma patients with Informed Consent Form
  2. Glioma patients with intact clinical information
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative Rapid Detection mutation of IDH, TERT and BRAF v600e | Intraoperative Rapid Detection mutation of IDH, TERT and BRAF v600e

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Huashan Hospital(West campus), Shanghai
  - Huashan Hospital, Shanghai
  - General Hospital of Ningxia Medical University, Yinchuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu J, Wu S, Cao D, Xiong Z, Zhang J, Zou Y, Wu Z, Nie Y, Luo C, Yao Y, Song Y, Jiao Y, Chen H, Ma H, Kang D, Mao Y, Yan H. Rapid diagnosis of adult-type diffuse glioma using a layered scheme. BMC Med. 2025 Jun 2;23(1):325. doi: 10.1186/s12916-025-04124-9. PMID 40457320